CLINICAL TRIAL: NCT03495726
Title: Mindfulness for Pain
Brief Title: Meditation for Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jennifer Mascaro, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00095434
Record Dates: First submitted 2018-04-02; First posted 2018-04-12 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pain
Keywords: Contemplative; Applications; Well-being
MeSH Terms: conditions — Chronic Pain | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Headspace app (Experimental): Participants randomized to use the mindfulness app for 6 weeks.
  Interventions: Behavioral: Headspace app
- Waitlist control group (No Intervention): This group will receive treatment as usual for 6 weeks. After the completing the 6-week surveys, the waitlist group will receive a subscription to the Headspace app.

INTERVENTIONS:
Behavioral: Headspace app — Headspace is a Contemplative Application (App) for Well-being (CAW). Participants will be provided initial instructions for downloading and using the Headspace app. The Headspace app includes guided meditations, articles and videos. Participants will be asked to engage in meditation practice for an average of 10 minutes a day during the 6-week training period.
  Other Names: Contemplative Applications for Well-being
  Arms: Headspace app

SUMMARY:
The general scope of the study involves meditation and its effects on pain management, narcotic use, and emotional well-being. Half of the participants will receive access to a meditation app, which they will be asked to use for at least 10 minutes every day for 6 weeks, while the other participants will be in the waitlist group and will receive a subscription to the meditation app after the 6 week study period ends. All participants will be asked to complete a set of questionnaires

DETAILED DESCRIPTION:
Chronic pain affects an estimated 11.2% of the US population, costs the United States approximately $635 billion per year in medical expenses and lost productivity, and fuels the current epidemic of opioid addiction. Understanding alternate approaches to chronic pain management is an imperative given new guidelines for the treatment of pain, and preliminary studies indicate that meditation programs may reduce the suffering and distress that accompanies chronic pain. However, much of the research on meditation for pain has examined the effects of scheduled group interventions, delivered in-person by instructors over the course of several weeks. Far less research has looked at the delivery method that is most common and arguably most sustainable for busy adults, namely, smart phone delivered Contemplative Applications (Apps) for Well-being (CAWs). The proposed study will examine the use and impact of a meditation apps in the context of pain. Participants will be randomized to either app or a wait-list group, and will be assessed in terms of self-reported pain, distress, narcotic use. To assess efficacy, the researchers will examine the longitudinal changes in all measures in the mindfulness app group, compared to wait-list control groups.

ELIGIBILITY:
Inclusion Criteria:

* Emory Healthcare patient

Exclusion Criteria:

* Non-english speaking patients
* Children, prisoners or other vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Change in Pain Catastrophizing Scale Score | Baseline, Week 3, Week 6, Week 14
  The Pain Catastrophizing Scale is a 13-item inventory that measures 3 elements of the perception of the intensity of pain (rumination, magnification, feeling helpless). Participants indicate the degree to which they agree with statements related their pain by selecting 0 = not at all, 1 = to a slight degree, 2 = to a moderate degree, 3 = to a great degree, 4 = all the time. There are three subscale scores assessing rumination, magnification and helplessness. All subscales are summed to produce a total score ranging from 0 to 52 with higher scores indicating the participant is having more thoughts about the pain they feel.
  helplessness. All subscales are summed to produce a total score ranging from 0 to 52 with higher scores indicating the participant is having more thoughts about the pain they feel.
Change in Brief Pain Inventory | Baseline, Week 3, Week 6, Week 14
  The Brief Pain Inventory is a 9-item inventory that measures both pain severity and pain interference in daily functioning with 2 scales. Questions are answered on an 11-point Likert scale from 0 to 10 and scales are scored by obtaining the mean for two separate scales: pain severity and pain interference.
Change in Current Opioid Misuse Measure (COMM) Score | Baseline, Week 3, Week 6, Week 14
  The COMM is a 17-item questionnaire assessing the aberrant medication-related behaviors of patients with chronic pain. Participants indicate how often they have experienced specific aberrant medication-related behaviors in the past 30 days on a scale from 0 (never) to 4 (very often). Total scores range from 0 to 68 with higher scores indicating more problematic behaviors.

SECONDARY OUTCOMES:
Change in Physical Functioning Subscale (PF-10) Score | Baseline, Week 3, Week 6, Week 14
  The PF-10 is a 10-item questionnaire assessing daily functioning. Participants respond to statements about how limited they are when performing daily living activities on a scale from 1 (cannot do) to 5 (not limited). Total scores range from 10 to 50 with higher scores indicating greater physical function.
Change in Basel Assessment of Adherence Immunosuppression Scale Score | Baseline, Week 3, Week 6, Week 14
  The Basel Assessment of Adherence Immunosuppression Scale is a 4-item questionnaire designed to assess adherence to medication regimen. Participants are asked about how well they have taken their medication during the past 4 weeks on a scale from 0 (never) to 5 (every day). Total scores range from 0 to 24 and higher score indicate greater problems with medication adherence.
Change in Depression Anxiety and Stress Scale (DASS) Score | Baseline, Week 3, Week 6, Week 14
  The Depression Anxiety and Stress Scale (DASS) is a 21-item survey asking about feelings of depression and anxiety that the respondent has experienced in the past week (for example, "I found myself getting upset at quite trivial things"). Respondents indicate the degree to which they agree with each statement on a scale of 0 to 3 where 0 = does not apply to me at all and 3 = applied to me very much, or most of the time. The depression subscale includes 14 items. A score of 0-9 indicates no depression, 10-13 indicates moderate depression, 14-20 is moderate depression, 21-27 is severe depression and scores of 28 and above indicate extremely severe depression.
Change in Brief Coping with Problems Experienced (COPE) Inventory | Baseline, Week 3, Week 6, Week 14
  The Brief COPE Inventory is a 28-item measurement assessing different types of coping mechanisms. Participants respond to statements expressing different ways to cope with life stress on a scale from 1 (I haven't been doing this at all) to 5 (I've been doing this a lot). This inventory is not designed for a summary score, rather, 14 separate scales with 2 items each can be examined and grouped into categories as desired. Total scores for each scale range from 2 to 10 with higher values indicating increased use of that coping mechanism.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Social Functioning - Short Form Score | Baseline, Week 3, Week 6, Week 14
  The PROMIS Social Functioning - Short Form is a 5-item measure assessing the ability to participate is social roles. Participants respond to statements about how their health impacts their social interactions on a scale from 1 (always) to 5 (never). Total scores range from 5 to 25 where higher scores indicate greater functioning in social roles.
Change in PROMIS Loneliness - Fixed Form Score | Baseline, Week 3, Week 6, Week 14
  The PROMIS Loneliness - Fixed Form is 5-item measure assessing loneliness. Participants report how often they have felt different aspects of loneliness on a scale from 1 (never) to 5 (always). Total scores range from 5 to 25 and higher scores indicate greater feelings of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mascaro, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided